CLINICAL TRIAL: NCT05007665
Title: Safety and Immune Response of COVID-19 Vaccination in Patients With Chronic Liver （CQMU）
Brief Title: Safety and Immune Response of COVID-19 Vaccination in Patients With Chronic Liver Diseases
Acronym: SIMPLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-48
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Liver Diseases; Covid19; Adverse Reaction to Vaccine
MeSH Terms: conditions — Liver Diseases; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Liver Diseases Patients/Healthy People: Chronic hepatitis (B OR C) , autoimmune hepatitis, liver cirrhosis, primary hepatocellular carcinoma
  Interventions: Biological: SARS-COV-2 VACCINE

INTERVENTIONS:
Biological: SARS-COV-2 VACCINE — the antibody titer and adverse reactions were observed.

SUMMARY:
On 11 February 2020, the International Committee for the Classification of Viruses named the disease caused by SAＲS-CoV-2 infection in humans as the new coronavirus pneumonia (coronavirus disease 2019, COVID-19). Due to the characteristics of liver microcirculation disturbance and immune function disorder in patients with chronic liver diseases (such as immune liver disease, chronic hepatitis C, liver cirrhosis, liver cancer, etc.), those patients has a higher risk of infection than the general population during the epidemic period. More attention should be paid to personal protection and disease prevention. Vaccination of COVID-19 vaccine can effectively prevent COVID-19 virus infection and delay or prevent patients from developing into critical illness and reduce mortality. To evaluate the safety and effectiveness of COVID-19 vaccine in those patients with chronic liver diseases, and to guide the COVID-19 vaccination more scientifically, reasonably and effectively, this study was carried out.

DETAILED DESCRIPTION:
Due to the characteristics of liver microcirculation disturbance and immune function disorder in patients with chronic liver diseases (such as autoimmune liver disease, chronic hepatitis C, liver cirrhosis, liver cancer, etc.), those patients has a higher risk of infection than the general population during the epidemic period. More attention should be paid to personal protection and disease prevention. Vaccination of COVID-19 / influenza vaccine can effectively prevent COVID-19 / influenza virus infection and delay or prevent patients from developing into critical illness and reduce mortality. The safety and effectiveness of COVID-19 / influenza vaccine in this population were evaluated in order to play a scientific and theoretical supporting role in guiding COVID-19 vaccination more scientifically, reasonably and effectively. The samples of this study were collected and tested in the second affiliated Hospital of Chongqing Medical University. Patients with contraindications for vaccination will be excluded. The detected indexes included blood routine test, liver function, COVID-19 antibody titer, antibody duration and other indexes of healthy people (control group) and patients with chronic liver disease before and after vaccination ( 1, 3, 6, 12 months after vaccination). The adverse reactions related to the vaccine were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy group were as follows: no history of hepatitis, no history of liver cirrhosis, no history of liver cancer and receiving the whole-course COVID-19 vaccination.
2. Patients with chronic liver disease diagnosed clinically or pathologically and receiving the whole-course COVID-19 vaccination.

Exclusion Criteria:

1. Patients previously diagnosed or with a history of contact with confirmed cases
2. Patients with contraindications for vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease vaccinated with SARS-Cov-2 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events after injection. | 4 weeks after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection. | 12 weeks after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection. | 24 weeks after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection. | 48 weeks after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.

SECONDARY OUTCOMES:
Titer and duration of COVID-19 antibody production after vaccination | 4 weeks after vaccination
  The titer and duration of COVID-19 antibody were produced at 4 weeks
Titer and duration of COVID-19 antibody production after vaccination | 12 weeks after vaccination
  The titer and duration of COVID-19 antibody were produced at 12 weeks
Titer and duration of COVID-19 antibody production after vaccination | 24 weeks after vaccination
  The titer and duration of COVID-19 antibody were produced at 24 weeks
Titer and duration of COVID-19 antibody production after vaccination | 48 weeks after vaccination
  The titer and duration of COVID-19 antibody were produced at 48 weeks after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with chronic liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, PH D, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The second affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Grohskopf LA, Alyanak E, Broder KR, Walter EB, Fry AM, Jernigan DB. Prevention and Control of Seasonal Influenza with Vaccines: Recommendations of the Advisory Committee on Immunization Practices - United States, 2019-20 Influenza Season. MMWR Recomm Rep. 2019 Aug 23;68(3):1-21. doi: 10.15585/mmwr.rr6803a1. PMID 31441906
- [Result] Xu X, Sun J, Nie S, Li H, Kong Y, Liang M, Hou J, Huang X, Li D, Ma T, Peng J, Gao S, Shao Y, Zhu H, Lau JY, Wang G, Xie C, Jiang L, Huang A, Yang Z, Zhang K, Hou FF. Seroprevalence of immunoglobulin M and G antibodies against SARS-CoV-2 in China. Nat Med. 2020 Aug;26(8):1193-1195. doi: 10.1038/s41591-020-0949-6. Epub 2020 Jun 5. PMID 32504052
- [Result] Shi Q, Hu Y, Peng B, Tang XJ, Wang W, Su K, Luo C, Wu B, Zhang F, Zhang Y, Anderson B, Zhong XN, Qiu JF, Yang CY, Huang AL. Effective control of SARS-CoV-2 transmission in Wanzhou, China. Nat Med. 2021 Jan;27(1):86-93. doi: 10.1038/s41591-020-01178-5. Epub 2020 Nov 30. PMID 33257893
- [Result] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Result] Long QX, Liu BZ, Deng HJ, Wu GC, Deng K, Chen YK, Liao P, Qiu JF, Lin Y, Cai XF, Wang DQ, Hu Y, Ren JH, Tang N, Xu YY, Yu LH, Mo Z, Gong F, Zhang XL, Tian WG, Hu L, Zhang XX, Xiang JL, Du HX, Liu HW, Lang CH, Luo XH, Wu SB, Cui XP, Zhou Z, Zhu MM, Wang J, Xue CJ, Li XF, Wang L, Li ZJ, Wang K, Niu CC, Yang QJ, Tang XJ, Zhang Y, Liu XM, Li JJ, Zhang DC, Zhang F, Liu P, Yuan J, Li Q, Hu JL, Chen J, Huang AL. Antibody responses to SARS-CoV-2 in patients with COVID-19. Nat Med. 2020 Jun;26(6):845-848. doi: 10.1038/s41591-020-0897-1. Epub 2020 Apr 29. PMID 32350462
- [Derived] Zhou Y, Chen Z, He Y, Peng X, Chang Y, Tan A, Li H, Cai D, Hu P, Chen M, Peng M, Xu H, Ren H. Humoral immune responses to inactivated COVID-19 vaccine up to 1 year in children with chronic hepatitis B infection. Front Cell Infect Microbiol. 2023 Jun 29;13:1201101. doi: 10.3389/fcimb.2023.1201101. eCollection 2023. PMID 37457966
- [Derived] Chen Z, Huang T, He T, Zha G, Zhu Q, Zhang G, Xiang D, Chen M, Li H, Ling N, Lan Y, Shi X, Zhang D, Xu P, Pan Q, Song R, Cao J, Zhang Y, Xiang H, Feng Y, Yang Z, Zhang B, Shen W, Cai D, Peng M, Hu P, Ren H. Humoral responses after primary and booster SARS-CoV-2 inactivated vaccination in patients with chronic hepatitis B virus infection: A longitudinal observational study. J Med Virol. 2023 Apr;95(4):e28695. doi: 10.1002/jmv.28695. PMID 36946505
- [Derived] He T, Ling N, Zhang G, Xiang D, Hu P, Peng M, Cai D, Zhang D, Chen M, Ren H. Decreased antibody response to influenza vaccine with an enhanced antibody response to subsequent SARS-CoV-2 vaccination in patients with chronic hepatitis B virus infection. Immun Inflamm Dis. 2023 Jan;11(1):e759. doi: 10.1002/iid3.759. PMID 36705404
- [Derived] He T, Zhou Y, Xu P, Ling N, Chen M, Huang T, Zhang B, Yang Z, Ao L, Li H, Chen Z, Zhang D, Shi X, Lei Y, Wang Z, Zeng W, Hu P, Lan Y, Zhou Z, Kang J, Huang Y, Shi T, Pan Q, Zhu Q, Ran X, Zhang Y, Song R, Xiang D, Xiao S, Zhang G, Shen W, Peng M, Cai D, Ren H. Safety and antibody response to inactivated COVID-19 vaccine in patients with chronic hepatitis B virus infection. Liver Int. 2022 Jun;42(6):1287-1296. doi: 10.1111/liv.15173. Epub 2022 Feb 28. PMID 35107848
- See also: World Health Organization (WHO) Influenza (Seasonal) 2018 Available from — http://who.int/en/news-room/fact-sheets/detail/influenza-(seasonal)